CLINICAL TRIAL: NCT05864521
Title: Effects of Nocturnal Inorganic Nitrate Supplementation on Physiological Function
Brief Title: Beetroot Juice and Sleep
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Joshua M. Bock, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 23-000874
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: Blood Pressure; Sleep

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Beetroot Juice Supplement (aBRJ) then Placebo Beetroot Juice Supplement (pBRJ) (Active Comparator): Subjects randomized to this arm of the study will have aBRJ administered during Visit 2 and then pBRJ administered during Visit 3.
  Interventions: Dietary Supplement: Active Beetroot Juice Supplement (aBRJ); Dietary Supplement: Placebo Beetroot Juice Supplement (pBRJ)
- Placebo Beetroot Juice Supplement (pBRJ) then Active Beetroot Juice Supplement (aBRJ) (Active Comparator): Subjects randomized to this arm of the study will have pBRJ administered during Visit 2 and then aBRJ administered during Visit 3.
  Interventions: Dietary Supplement: Active Beetroot Juice Supplement (aBRJ); Dietary Supplement: Placebo Beetroot Juice Supplement (pBRJ)

INTERVENTIONS:
Dietary Supplement: Active Beetroot Juice Supplement (aBRJ) — aBRJ will consist of 70ml concentrated beetroot juice with 6.45-7.26mmol inorganic nitrate (range for inter-batch variability) taken orally.
Dietary Supplement: Placebo Beetroot Juice Supplement (pBRJ) — pBRJ will consist of 70ml concentrated beetroot juice and will be chemically devoid of inorganic nitrate taken orally.

SUMMARY:
The purpose of this study is to investigate the effects of acute inorganic nitrate supplementation (with beetroot) on the regulation of sleep and neurovascular physiology.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 or 65-80 years of age

Exclusion Criteria:

* Coronary artery disease
* Heart failure
* Pregnancy
* Diabetes
* Sleep disorders
* Shift workers
* Individuals who typically go to sleep after midnight
* Individuals who traveled across ≥2 time zones within one week of study visits
* Individuals with a history frequent kidney stones
* BMI ≥35.0kg/m2
* Use of nicotine-containing products within the two years preceding study visits
* Use of allopurinol, proton pump inhibitors, or other medications/supplements which interfere with the nitrate-nitrite-nitric oxide pathway or outcome measures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in the amount of time in stage three sleep | Baseline, approximately 30 days, and approximately 60 days
  Measured overnight polysomnography (PSG) used to identify sleep staging, reported in minutes
Change in sleep quality | Baseline, approximately 30 days, and approximately 60 days
  Measured by Pittsburgh Sleep Quality Index which measures the severity of sleep disturbances. Possible scores range from 0 to 21 with higher scores indicating a worse outcome/more severe symptoms of sleep disturbance.
Change in self-reported sleep quality | Baseline, approximately 30 days, and approximately 60 days
  Measured on a visual analog scale of 1-10, where 1 is not at all sleepy and 10 is as sleepy as you can imagine, how sleepy are you right now?
Change in sleepiness | Baseline, approximately 30 days, and approximately 60 days
  Measured by the Stanford Sleepiness Scale that asks participate to rank their degree of sleepiness where 1 would indicate the subject currently feels least sleepy and 7 would indicate the subject feels the most sleepy.
Change in daytime sleepiness | Baseline, approximately 30 days, and approximately 60 days
  Measured by Epworth Sleepiness Scale. The test is a list of eight situations in which you rate your tendency to become sleepy on a scale of 0, no chance of dozing, to 3, high chance of dozing. Total score is graded from 0-24. 0-7:It is unlikely that you are abnormally sleepy. 8-9:You have an average amount of daytime sleepiness. 10-15:You may be excessively sleepy depending on the situation. You may want to consider seeking medical attention. 16-24:You are excessively sleepy and should consider seeking medical attention.

SECONDARY OUTCOMES:
Change in blood pressure | Baseline, approximately 30 days, and approximately 60 days
  Measured in millimeters of mercury (mmHg)
Change in sympathetic nerve burst frequency | Baseline, approximately 30 days, and approximately 60 days
  Measured by Microneurography reported as number of nerve bursts per minute (burst/min)
Change in sympathetic nerve burst incidence | Baseline, approximately 30 days, and approximately 60 days
  Measured by Microneurography reported as number of nerve burst per 100 heart beats (burst/100 heart beats)
Change in sympathetic nerve burst amplitude (AU) | Baseline, approximately 30 days, and approximately 60 days
  Measured by Microneurography reported in arbitrary units (AU)
Change in total muscle sympathetic nerve activity (MSNA) | Baseline, approximately 30 days, and approximately 60 days
  Measured by Microneurography reported burst arbitrary units per minute (AU/min)
Change in arterial stiffness | Baseline, approximately 30 days, and approximately 60 days
  Measured by applanation tonometry reported as aortic pulse wave velocity (m/sec)
Change in endothelial function | Baseline, approximately 30 days, and approximately 60 days
  Ultrasound assessment of flow-mediated vasodilation of the brachial artery. Brachial artery diameter and blood velocity will be measured after deflation to measure endothelial function.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Bock, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No